CLINICAL TRIAL: NCT03535571
Title: A Proof-of-concept Study to Evaluate the Efficacy of Salmon Protein Hydrolysate Powder on Energy Increase and Anti-inflammatory Modulation in Healthy Males and Females
Brief Title: A Study to Evaluate the Efficacy of Salmon Protein Hydrolysate Powder on Energy Increase and Anti-inflammatory Modulation in Healthy Males and Females
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hofseth Biocare ASA (Industry)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 18PEHH
Record Dates: First submitted 2018-05-14; First posted 2018-05-24 (Actual); Results first posted 2019-08-19 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-07

CONDITIONS: Healthy
Keywords: Energy increase; Energy; Healthy; anti-inflammatory; Open-label; Salmon protein; Natural health product; Dietary supplement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Salmon Protein Hydrolysate (CollaGo®) (Experimental): Dose: 1 sachet of CollaGo® will be mixed with 100-300 mL of water and consumed daily at breakfast.
  Interventions: Dietary Supplement: Salmon Protein Hydrolysate

INTERVENTIONS:
Dietary Supplement: Salmon Protein Hydrolysate — 4g of salmon protein hydrolysate per serving.
  Other Names: CollaGo®

SUMMARY:
The objective of this study is to evaluate the efficacy of Salmon Protein Hydrolysate Powder (CollaGo®) on energy increase and anti-inflammatory modulation in healthy males and females. Eligible participants will be asked to consume 1 sachet of CollaGo for 128 days and keep a study diary. Assessments will be measured at the randomization visit, and the end of study visit.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female, 30-60 years of age
2. Female participant is not of child bearing potential, defined as females who have had a hysterectomy or oophorectomy, bilateral tubal ligation or are post-menopausal (natural or surgically with > 1 year since last menstruation) or,

   Females of childbearing potential must agree to use a medically approved method of birth control and have a negative urine pregnancy test result. All hormonal birth control must have been in use for a minimum of three months. Acceptable methods of birth control include:
   * Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)
   * Double-barrier method
   * Intrauterine devices
   * Non-heterosexual lifestyle or agrees to use contraception if planning on changing to heterosexual partner(s)
   * Vasectomy of partner (shown successful as per appropriate follow-up)
3. BMI of 18.5 kg/m²-32.5 kg/m²
4. Agrees to comply with study procedures
5. Willing to commit to taking product for 128 days
6. Agrees to provide voluntary, written, informed consent to participate in the study
7. Agrees to maintain normal diet and exercise routine throughout the study
8. Healthy as determined by medical history, medical physical test for good health, and laboratory results

Exclusion Criteria:

1. Women who are pregnant, breastfeeding, or planning to become pregnant during the trial
2. Blood donation during or within 30 days of the last study visit
3. Taking any specific energy supplements or vitamins at least 1 month prior to and during the trial as assessed by the QI
4. Unstable weight for the last 2 months prior to the study assessed case by case by QI
5. Individuals on a low protein diet
6. Excessive consumption of alcohol equivalent to >2 alcoholic drinks/day
7. Use of marijuana assessed case by case by QI
8. Known allergy to the test material's active or inactive ingredients
9. Clinically significant abnormal Physical Examination results at screening
10. Participation in clinical trials in the past 30 days
11. Cognitively impaired and/or unable to give informed consent
12. current cardiovascular disorders or uncontrolled blood pressure will be assessed by QI)
13. Verbal confirmation of history of or current diagnosis of bleeding/blood disorder
14. Verbal confirmation of Type I or Type II diabetes
15. Verbal confirmation of kidney disease
16. Verbal confirmation of history of liver disease
17. Anemia based on hemoglobin and hematocrit at screening
18. Thyroid disease assessed case by case by QI
19. Iron Supplementation
20. Mood stabilizers assessed case by case by QI
21. Energy boosting supplements
22. Individuals on workout supplements
23. Habitual users of energy drinks
24. Melatonin supplementation assessed case by case by QI
25. Autoimmune disease or if immune-compromised (i.e. HIV positive, use of anti-rejection medication, rheumatoid arthritis, Hepatitis B/C positive)
26. Surgical procedures which may impact the study outcomes within the past 3 months to be assessed by the QI
27. Cancer, except skin cancers completely excised with no chemotherapy or radiation with a follow up that is negative. Volunteers with cancer in full remission will be assessed by the QI for inclusion.
28. Presence or history of neurological disorders or significant psychiatric illness as assessed by QI
29. Any other condition, in the QI's opinion, which may adversely affect the participant's ability to complete the study or its measures or which may pose significant risk to the participant

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-06-05 (Actual); Primary Completion 2018-10-23 (Actual); Study Completion 2018-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Crowley, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Science Inc., London, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Salmon Protein Hydrolysate (CollaGo): Dose: 1 sachet of CollaGo will be mixed with 100-300 mL of water and consumed daily at breakfast.
  Salmon Protein Hydrolysate: 4g of salmon protein hydrolysate per serving.
Period: Overall Study
Arm/Group | Salmon Protein Hydrolysate (CollaGo)
Started | 20
Completed | 19
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Salmon Protein Hydrolysate (CollaGo)
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.45 (5.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African or African American | 2
  East Asian or South East Asian | 3
  Hispanic or Latino | 1
  South American | 3
  Western or Eastern European White | 10
  Native American | 1

OUTCOME MEASURES:

1. Primary Outcome: The Change From Baseline (Day 0) to End-of-study (Day 128) in Energy Level After a 128-day Supplementation With Collagenic Salmon Protein Hydrolysate Powder (CollaGo®)
Description: This questionnaire consists of a total of 30 questions that assess vitality and quality of life. The responses for these questions range from 1 to 7, where 1 indicates "never" or "not at all true" 4 indicates "sometimes" or "somewhat true" and 7 indicates "always" or "very true" depending on the item that is assessed by the question.
  15 of the 30 questions are positively keyed in which a higher score indicates a better outcome and remaining 15 questions are negatively keyed where a lower score indicates a better outcome. The responses on the negatively keyed questions will be reversed prior to calculating the total score (i.e. a response of 1 will be considered as 7, 2 will be considered as 6, etc.). Total range will be 30-210, where a higher total score indicates a better outcome and a lower total score indicates a worse outcome.
Time Frame: Baseline (Day 0) to end-of-study (Day 128)
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Salmon Protein Hydrolysate (CollaGo®)
Number analyzed (Participants) | 19
score on a scale | 13.89 (20.49)

2. Secondary Outcome: Change From Baseline to Day 128 in Red Blood Cell (RBC) Count After Supplementation With Collagenic Salmon Protein Hydrolysate Powder (CollaGo®)
Time Frame: Baseline (Day 0) to end-of-study (Day 128)
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: cells x10^12/L
Groups:
- Salmon Protein Hydrolysate (CollaGo): Dose: 1 sachet of CollaGo® will be mixed with 100-300 mL of water and consumed daily at breakfast.
  Salmon Protein Hydrolysate: 4g of salmon protein hydrolysate per serving.
Arm/Group | Salmon Protein Hydrolysate (CollaGo)
Number analyzed (Participants) | 20
cells x10^12/L | 0.08 (0.23)

3. Secondary Outcome: Change From Baseline to Day 128 in Mean Corpuscular Volume (MCV) After Supplementation With Collagenic Salmon Protein Hydrolysate Powder (CollaGo®)
Time Frame: Baseline (Day 0) to end-of-study (Day 128)
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: fL
Arm/Group | Salmon Protein Hydrolysate (CollaGo®)
Number analyzed (Participants) | 20
fL | -1.1 (2.36)

4. Secondary Outcome: Change From Baseline to Day 128 in Mean Corpuscular Hemoglobin (MCH) After Supplementation With Collagenic Salmon Protein Hydrolysate Powder (CollaGo®)
Time Frame: Baseline (Day 0) to end-of-study (Day 128)
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: pg
Arm/Group | Salmon Protein Hydrolysate (CollaGo®)
Number analyzed (Participants) | 20
pg | 0.09 (0.77)

5. Secondary Outcome: Change From Baseline to Day 128 in Mean Corpuscular Hemoglobin Concentration (MCHC) After Supplementation With Collagenic Salmon Protein Hydrolysate Powder (CollaGo®)
Time Frame: Baseline (Day 0) to end-of-study (Day 128)
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Salmon Protein Hydrolysate (CollaGo®)
Number analyzed (Participants) | 20
g/L | 4.65 (12.9)

6. Secondary Outcome: Change From Baseline to Day 128 in Hematocrit After Supplementation With Collagenic Salmon Protein Hydrolysate Powder (CollaGo®)
Time Frame: Baseline (Day 0) to end-of-study (Day 128)
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: L/L
Arm/Group | Salmon Protein Hydrolysate (CollaGo®)
Number analyzed (Participants) | 20
L/L | 0 (0.02)

7. Secondary Outcome: Change From Baseline to Day 128 in Red Cell Distribution Width (RDW) After Supplementation With Collagenic Salmon Protein Hydrolysate Powder (CollaGo®)
Time Frame: Baseline (Day 0) to end-of-study (Day 128)
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: percent change in size
Arm/Group | Salmon Protein Hydrolysate (CollaGo®)
Number analyzed (Participants) | 20
percent change in size | -0.79 (0.51)

8. Secondary Outcome: Change From Baseline to Day 128 in Hemoglobin (Hb) After Supplementation With Collagenic Salmon Protein Hydrolysate Powder (CollaGo®)
Time Frame: Baseline (Day 0) to end-of-study (Day 128)
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Salmon Protein Hydrolysate (CollaGo®)
Number analyzed (Participants) | 20
g/L | 3 (7.41)

9. Secondary Outcome: Change From Baseline to Day 128 in Relative Expression of 84 Stress Genes After Supplementation With Collagenic Salmon Protein Hydrolysate Powder (CollaGo®)
Description: Evaluated by oxidative stress-related gene RT Profiler PCR array. Seven of the 84 genes were upregulated, which are highlighted in the results.
Time Frame: Baseline (Day 0) to end-of-study (Day 128)
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: Fold change
Arm/Group | Salmon Protein Hydrolysate (CollaGo®)
Number analyzed (Participants) | 20
Fold change
  APOE | 2.60 (0.21)
  FTH1 | 3.73 (0.40)
  GCLC | 2.64 (0.35)
  GPX1 | 2.96 (0.29)
  HMOX1 | 4.10 (0.23)
  NQO1 | 3.12 (0.17)
  SOD1 | 3.06 (0.19)

10. Secondary Outcome: Change From Baseline to Day 128 in Total Reactive Oxygen Species/Reactive Nitrogen Species Free Radical Activity After Supplementation With Collagenic Salmon Protein Hydrolysate Powder (CollaGo®)
Description: Assessed by ROS/RNS assay
Time Frame: Baseline (Day 0) to end-of-study (Day 128)
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Salmon Protein Hydrolysate (CollaGo®)
Number analyzed (Participants) | 20
mmol/L | -0.14 (0.11)

11. Secondary Outcome: Change From Baseline to Day 128 in Levels of Human Inflammatory Cytokine IL-1 Alpha After Supplementation With Collagenic Salmon Protein Hydrolysate Powder (CollaGo®).
Description: Measured by the Multi-Analyte ELISArray
Time Frame: Baseline (Day 0) to end-of-study (Day 128)
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Salmon Protein Hydrolysate (CollaGo®)
Number analyzed (Participants) | 20
pg/mL | 0.01 (0.05)

12. Secondary Outcome: Change From Baseline to Day 128 in Levels of Human Inflammatory Cytokine IL-4 After Supplementation With Collagenic Salmon Protein Hydrolysate Powder (CollaGo®).
Description: Measured by the Multi-Analyte ELISArray
Time Frame: Baseline (Day 0) to end-of-study (Day 128)
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Salmon Protein Hydrolysate (CollaGo®)
Number analyzed (Participants) | 20
pg/mL | 0 (0.03)

13. Secondary Outcome: Change From Baseline to Day 128 in Levels of Human Inflammatory Cytokine IL-6 After Supplementation With Collagenic Salmon Protein Hydrolysate Powder (CollaGo®).
Description: Measured by the Multi-Analyte ELISArray
Time Frame: Baseline (Day 0) to end-of-study (Day 128)
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Salmon Protein Hydrolysate (CollaGo®)
Number analyzed (Participants) | 20
pg/mL | -0.07 (0.28)

14. Secondary Outcome: Change From Baseline to Day 128 in Levels of Human Inflammatory Cytokine IL-10 After Supplementation With Collagenic Salmon Protein Hydrolysate Powder (CollaGo®).
Description: Measured by the Multi-Analyte ELISArray
Time Frame: Baseline (Day 0) to end-of-study (Day 128)
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Salmon Protein Hydrolysate (CollaGo®)
Number analyzed (Participants) | 20
pg/mL | 1.39 (0.98)

15. Secondary Outcome: Change From Baseline to Day 128 in Levels of Human Inflammatory Cytokine IL-11 After Supplementation With Collagenic Salmon Protein Hydrolysate Powder (CollaGo®).
Description: Measured by the Multi-Analyte ELISArray.
Time Frame: Baseline (Day 0) to end-of-study (Day 128)
Population: This measure was not included in the Multi-Analyte ELISArray analysis, therefore there is no data to report.
Arm/Group | Salmon Protein Hydrolysate (CollaGo)
Number analyzed (Participants) | 0

16. Secondary Outcome: Change From Baseline to Day 128 in Levels of Human Inflammatory Cytokine IL-13 After Supplementation With Collagenic Salmon Protein Hydrolysate Powder (CollaGo®).
Description: Measured by the Multi-Analyte ELISArray
Time Frame: Baseline (Day 0) to end-of-study (Day 128)
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Salmon Protein Hydrolysate (CollaGo®)
Number analyzed (Participants) | 20
pg/mL | -0.14 (1.29)

17. Secondary Outcome: Change From Baseline to Day 128 in Levels of Human Inflammatory Cytokine TGF-Beta After Supplementation With Collagenic Salmon Protein Hydrolysate Powder (CollaGo®)
Description: Measured by the Multi-Analyte ELISArray
Time Frame: Baseline (Day 0) to end-of-study (Day 128)
Population: This measure was not included in the Multi-Analyte ELISArray analysis, therefore there is no data to report.
Arm/Group | Salmon Protein Hydrolysate (CollaGo)
Number analyzed (Participants) | 0

18. Secondary Outcome: Change From Baseline to Day 128 in Glycated Hemoglobin (HbA1c) After Supplementation With Collagenic Salmon Protein Hydrolysate Powder (CollaGo®)
Time Frame: Baseline (Day 0) to end-of-study (Day 128)
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: percentage of glucose bound to RBCs
Arm/Group | Salmon Protein Hydrolysate (CollaGo®)
Number analyzed (Participants) | 20
percentage of glucose bound to RBCs | 0.08 (0.17)

19. Secondary Outcome: Change From Baseline to Day 128 in Fasting Glucose After Supplementation With Collagenic Salmon Protein Hydrolysate Powder (CollaGo®)
Time Frame: Baseline (Day 0) to end-of-study (Day 128)
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Salmon Protein Hydrolysate (CollaGo®)
Number analyzed (Participants) | 20
mmol/L | -0.15 (0.45)

20. Secondary Outcome: Change in Score of the Hair, Nails, and Skin Self-Assessment Questionnaire After 128-day Supplementation With Collagenic Salmon Protein Hydrolysate Powder (CollaGo®)
Description: This questionnaire consists of a total of 7 questions that assess the participant's perception on hair (4 questions), nail (1 question) and skin health (2 question). The response to each question can range from 1 to 6 where 1 indicates "greatly satisfied" and 6 indicates "greatly dissatisfied".
  The range for the total score on this questionnaire is 7-42. Lower total score indicates a better outcome, and higher total score indicates a worse outcome.
Time Frame: Baseline (Day 0) to end-of-study (Day 128)
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Salmon Protein Hydrolysate (CollaGo®)
Number analyzed (Participants) | 19
score on a scale | -0.74 (1.22)

21. Other Pre Specified Outcome: The Incidence of Adverse Events Following a 128-day Supplementation
Time Frame: Baseline (Day 0) to end-of-study (Day 128)
Population: Frequency Threshold for Reporting Other Adverse Events: 5%. Full information can be found in the adverse events section. Summary can be found below.
Measure: Count of Participants; unit: Participants
Arm/Group | Salmon Protein Hydrolysate (CollaGo)
Number analyzed (Participants) | 20
Participants | 6

22. Other Pre Specified Outcome: The Effect of a 128-day Supplementation on Weight
Time Frame: Baseline (Day 0) to end-of-study (Day 128)
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Salmon Protein Hydrolysate (CollaGo®)
Number analyzed (Participants) | 20
kg | 0.34 (2.02)

23. Other Pre Specified Outcome: The Effect of a 128-day Supplementation on Blood Pressure
Time Frame: Baseline (Day 0) to end-of-study (Day 128)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Salmon Protein Hydrolysate (CollaGo)
Number analyzed (Participants) | 20
mmHg
  Systolic Blood Pressure | 4.37 (8.01)
  Diastolic Blood Pressure | 0.48 (7.25)

24. Other Pre Specified Outcome: The Effect of a 128-day Supplementation on Heart Rate
Time Frame: Baseline (Day 0) to end-of-study (Day 128)
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Salmon Protein Hydrolysate (CollaGo®)
Number analyzed (Participants) | 20
beats per minute | -0.35 (16.61)

25. Other Pre Specified Outcome: The Effect of a 128-day Supplementation on Waist Circumference
Time Frame: Baseline (Day 0) to end-of-study (Day 128)
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Salmon Protein Hydrolysate (CollaGo®)
Number analyzed (Participants) | 20
cm | 0.86 (5.8)

26. Other Pre Specified Outcome: The Effect of a 128-day Supplementation on Hip Circumference
Time Frame: Baseline (Day 0) to end-of-study (Day 128)
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Salmon Protein Hydrolysate (CollaGo®)
Number analyzed (Participants) | 20
cm | -0.48 (2.1)

ADVERSE EVENTS:
Time Frame: 128-days
Arm/Group | Salmon Protein Hydrolysate (CollaGo)
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 1/20
Other Adverse Events (participants affected / at risk) | 5/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Salmon Protein Hydrolysate (CollaGo) (N=20)
Mental breakdown (Psychiatric disorders) | 1 (1) — Determined to not be related to the study product
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Salmon Protein Hydrolysate (CollaGo) (N=20)
Back, muscle, leg pain (Musculoskeletal and connective tissue disorders) | 2 (4)
Neuropathy, paresthesia, tension headache (Nervous system disorders) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study was conducted by a contract research organization (CRO) of which the PI is a contract employee. The agreement between the CRO and sponsor indicates that all rights to discuss and publish the trial results belong to the sponsor.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-03): https://cdn.clinicaltrials.gov/large-docs/71/NCT03535571/Prot_SAP_000.pdf